CLINICAL TRIAL: NCT04925947
Title: Phase II Study of KN046 in Patients With Thymic Carcinoma Who Failed Immune Checkpoint Inhibitors
Brief Title: A Study of KN046 in Patients With Thymic Carcinoma Who Failed Immune Checkpoint Inhibitors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data collected did not support the study endpoints
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022493
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Thymic Carcinoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KN046 (Experimental): KN046 will be given intravenously every 2 weeks.
  Interventions: Drug: KN046

INTERVENTIONS:
Drug: KN046 — KN046 will be given intravenously at 5 mg/kg every 2 weeks. A cycle is defined as 2 treatments (28 days). Treatment will be given until progression, excessive toxicity, or up to two years.

SUMMARY:
This study will assess the safety and efficacy of the study drug KN046 in patients with advanced thymic carcinoma who progressed after prior treatment with immune checkpoint inhibitor therapy.

DETAILED DESCRIPTION:
Patients will receive KN046 intravenously at 5 mg/kg every 2 weeks until progression or excessive toxicity for up to to two years, with the goal of this trial to contribute to the development of active and well tolerated treatments for patients who have progressed on prior treatment therapies.

Recently, molecules that combine PD-1 and CTLA-4 have been developed for patients with lung cancer, with the hope that targeted therapy will be more effective than standard of care therapies. KN046 is believed to be less toxic than other targeted therapies with an assumption that the whole molecule can actively target tumor tissue for a much higher affinity of the anti-PD-L1 portion and a weaker affinity for anti-CTLA-4, leading to less autoimmune disorders and toxicities for patients than seen with other targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Male or female, 18 years of age or older; willing and able to complete all required procedures of study.
* Pathologically confirmed diagnosis of thymic carcinoma; a tumor sample is required for confirmation of pathological diagnosis and further studies on the tumor tissue.
* Inoperable or metastatic disease.
* Progressive disease documented in the last 6 months.
* Has failed platinum-based chemotherapy, with progression either during or after treatment.
* Had failed at least one regimen of systemic therapy containing immune checkpoint blockade therapy targeting PD-1, PD-L1, or CTLA-4 for locally advanced unresectable or metastatic disease. Subjects should have documented progressive disease while or after an immune checkpoint therapy. If subjects discontinued therapy due to reasons other than progressive disease, subjects should have completed at least 2 cycles of immune checkpoint therapy.
* Baseline measurable disease according to RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* ECOG performance status of 0 or 1.
* Adequate organ function assessed within 7 days prior to first trial treatment:

Hematological function:

ANC≥1.5 x 109/L; Hemoglobin≥9 g/dL; Platelets≥100 x 109/L

Renal function:

Calculated creatinine clearance≥60 mL/min (Cockcroft-Gault method)

Hepatic function:

Total bilirubin≤1.5 x ULN (or 2.5 x ULN for documented Gilberts' syndrome); ALT/AST≤3.0 x ULN (or 5.0 x ULN for documented liver metastasis); INR or aPTT ≤1.5 x ULN

* Have a life expectancy of at least 3 months.
* If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment.
* If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

* Thymomas, thymolipoma, germ cell tumors, teratomas, seminomas.
* Leptomeningeal metastasis or untreated active CNS metastasis or leptomeningeal metastasis. Subjects with CNS metastasis may be eligible provided they are treated and clinically stable for at least 4 weeks and have no evidence of new or enlarging brain metastases and also are off steroids 7 days prior to first trial treatment.
* Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter, prior to the first dose of trial treatment.
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment.
* Radiation within 4 weeks prior to the first administration of trial treatment; palliative radiation will be allowed if more than 2 weeks before start of KN046 treatment.
* Subjects receiving immunosuppressive agents (such as systemic steroids); topical use of steroids and steroid inhalers are allowed. Replacement therapy because of adrenal insufficiency is also allowed.
* Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines).
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
* History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent, including but not limited to:

Myasthenia gravis (MG), Good syndromes, ISAACS syndromes, polymyositis, myocarditis, neuromuscular syndrome (myotonic dystrophy myositis, Eaton-Lambert syndrome), blood disorders (red cell aplasia, hypogammaglobulinemia, T-cell deficiency syndrome, erythrocytosis, pancytopenia, megakaryocytopenia, T-cell lymphocytosis, pernicious anemia), systemic lupus erythematosus, sarcoidosis, scleroderma, Crohn's disease, inflammatory bowel disease, Wegener syndrome (granulomatosis with polyangitis, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis), autoimmune hepatitis, systemic sclerosis (for example scleroderma), Hashimoto thyroiditis (with the exception as stated below), hyperparathyroidism, stiff-person syndrome, Addison disease, panhypopituitarism, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome) etc.

NOTE: Subjects with Type I diabetes, vitiligo, psoriasis, hypo- or hyperthyroid disease, Sjögren syndrome not requiring immunosuppressive treatment are eligible. Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤10 mg or equivalent prednisone per day. Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intra-ocular, or inhalation) are acceptable.

* Previous malignant disease other than the target malignancy to be investigated in this study with the exception of adequately treated non-melanomatous cancers of the skin, in situ carcinoma of the prostate/cervical/breast cancer, or other malignancy treated at least 5 years previously with surgery and/or curative radiotherapy, and there is no evidence of recurrence since that time.
* History of uncontrolled intercurrent illness including but not limited to: Active HBV or HCV infection (If HBsAg and HCV antibody positive, HBV DNA and HCV RNA assay should be performed. Subjects may be eligible if HBV DNA ≤ 500 UI/ml (or 2000 copies/ml) or HCV RNA negative); Known HIV infection or known history of acquired immune deficiency syndrome (AIDS); Active tuberculosis infection; Active infection within 2 weeks prior to the first dose of trial treatment that require the use of systemic antibiotics; Hypertension uncontrolled by standard therapies (not stabilized to 150/90 mmHg); Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), myocardial infarction (< 6 months prior to enrolment), unstable angina pectoris, congestive heart failure (New York Heart Association Classification Class II-IV) or serious cardiac arrhythmia requiring medication (including corrected QT interval prolongation of > 470 msec calculated according to Fridericia and/or pacemaker or prior diagnosis of congenital long QT syndrome
* Persisting toxicity related to prior therapy (including any prior investigational therapy) of CTCAE ≥ grade 2 (NCI-CTCAE v5.0) or related toxicity not recovery to baseline, with the exception of alopecia of any grade.
* Prior allo-HSCT or solid organ transplant.
* Known severe hypersensitivity reactions to antibody drug (≥ grade 3 NCI-CTCAE v5.0), any history of anaphylaxis, uncontrolled asthma (that is, 3 or more features of partially controlled asthma), or any history of severe drug hypersensitivity (for example immune mediated liver toxicity, immune mediated thrombocytopenia or anemia).
* Is pregnant or breastfeeding.
* Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance. These include but are not limited to psychiatric or substance abuse disorder, moderate to large pleural fluid/cardiac effusion/ascites, or recurrent/refractory pleural fluid/cardiac effusion/ascites.
* .Subjects with history or baseline positive antiacetylcholine receptor (AChR) autoantibody and anti-MuSK autoantibody.
* Subjects who developed grade 3 or above immune related AE which could not be managed by steroid or immune suppressant will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ma, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KN046
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | KN046
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Anti-tumor Activity of KN046 in Subjects With Thymic Carcinoma, Determined by Subject Disease Response Rate Defined by the RECIST 1.1 Criteria.
Description: Disease response rate
Time Frame: Up to 8 weeks
Measure: Number; unit: count of participants
Arm/Group | KN046
Number analyzed (Participants) | 4
count of participants | 0

2. Secondary Outcome: Safety of KN046 in Subjects With Thymic Carcinoma, Measured by the Number of Adverse Events That Occur in Subjects While Receiving Study Treatment.
Time Frame: Up to 8 weeks
Measure: Number; unit: adverse events
Arm/Group | KN046
Number analyzed (Participants) | 4
adverse events | 20

3. Secondary Outcome: Tolerability of KN046 in Subjects With Thymic Carcinoma, Measured by the Severity of Adverse Events That Occur in Subjects While Receiving Study Treatment, Assessed Using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Description: AEs are graded using the following criteria using Common Terminology Criteria for Adverse events v5.0:
  Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death related to AE.
Time Frame: Up to 8 weeks
Measure: Number; unit: adverse events
Arm/Group | KN046
Number analyzed (Participants) | 4
adverse events
  Grade 1 | 13
  Grade 2 | 7
  Grade 3 | 6
  Grade 4 | 1

4. Secondary Outcome: Duration of Response for KN046 in Subjects With Thymic Carcinoma, Determined by Subject Disease Response Rate Defined by the RECIST 1.1 Criteria.
Time Frame: Up to 8 weeks
Measure: Number; unit: months
Arm/Group | KN046
Number analyzed (Participants) | 4
months | 0

5. Secondary Outcome: Progression Free Survival (PFS) for KN046 in Subjects With Thymic Carcinoma, Determined by Subject Disease Response Rate Defined by the RECIST 1.1 Criteria.
Time Frame: Up to 8 weeks
Measure: Number; unit: participants
Arm/Group | KN046
Number analyzed (Participants) | 4
participants | 0

6. Secondary Outcome: Overall Survival (OS) for KN046 in Subjects With Thymic Carcinoma, Determined by Subject Disease Response Rate Defined by the RECIST 1.1 Criteria.
Time Frame: Up to 8 weeks
Measure: Number; unit: participants
Arm/Group | KN046
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: Up to 11.5 weeks
Description: Expected adverse events to monitor include infusion-related adverse events, hypersensitivity reactions and immune-related adverse events.
Arm/Group | KN046
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KN046 (N=4)
Absolute Lymphocyte Count Decreased (Investigations) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KN046 (N=4)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chest pain - Cardiac (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early and participant enrollment was low, resulting in a small sample size (N=4). Having a small sample size may reduce statistical reliability and generalizability of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/47/NCT04925947/Prot_SAP_000.pdf